CLINICAL TRIAL: NCT04668989
Title: Evaluation of the Performance of Different Daily Disposable Lens Designs in Habitual Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-118
Record Dates: First submitted 2020-12-04; First posted 2020-12-16 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- stenfilcon A - (Test lens) (Experimental): Subjects will be randomized to wear test lenses for one week then cross-over to the control lenses for one week.
  Interventions: Device: stenfilcon A - (Test lens); Device: kalifilcon A - (Control Lens)
- kalifilcon A - (Control Lens) (Active Comparator): Subjects will be randomized to wear control lenses for one week then cross-over to the test lenses for one week.
  Interventions: Device: stenfilcon A - (Test lens); Device: kalifilcon A - (Control Lens)

INTERVENTIONS:
Device: stenfilcon A - (Test lens) — Subjects will be randomized to wear test lenses for one week.
Device: kalifilcon A - (Control Lens) — Subjects will be randomized to wear control lenses for one week.

SUMMARY:
The main objective of the study is to refit existing soft lens wearers with two different daily disposable contact lens types, Lens A and Lens B, to determine their performance after one week of wear.

DETAILED DESCRIPTION:
This study is a prospective, bilateral eye, double-masked, randomized, 1-week cross-over, daily-wear design involving two different daily disposable lens types. Each lens type will be worn for approximately one week, during which participants record their subjective lens-wear experience.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Self reports having a full eye examination in the previous two years;
4. Anticipates being able to wear the study lenses for at least 8 hours a day, 7 days a week;
5. Is willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wears soft contact lenses, for the past 3 months minimum;
7. Has refractive astigmatism no higher than -0.75DC in each eye;
8. Can be fit and achieve binocular distance vision of at least 20/30 Snellen (Available lens parameters are sphere -1.00 to -6.00D, 0.25D steps).

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Habitually wears one of the study contact lenses;
3. Has any known active* ocular disease and/or infection that contraindicates contact lens wear;
4. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
5. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
6. Has known sensitivity to the diagnostic sodium fluorescein used in the study;
7. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
8. Has undergone refractive error surgery or intraocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Study Director — Centre for Ocular Research & Education
Locations (4):
- United States (4):
  - Complete Eye Care of Medina, Medina, Minnesota
  - Sacco Eye Group, PLLC, Vestal, New York
  - Athens Eye Care, Athens, Ohio
  - Nittany Eye Associates, College, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 68 participants were screened, 2 subjects discontinued, and 66 subjects were dispensed with the study lenses.
Groups:
- Stenfilcon A - (Test Lens) Then Kalifilcon A (Control Lens): Subjects were randomized to wear test lenses for one week then cross-over to the control lenses for one week.
  stenfilcon A - (Test lens)
  kalifilcon A - (Control lens)
- Kalifilcon A - (Control Lens) Then Stenfilcon A - (Test Lens): Subjects were randomized to wear control lenses for one week then cross-over to the test lenses for one week.
  stenfilcon A - (Test lens)
  kalifilcon A - (Control Lens)
Period: First Intervention
Arm/Group | Stenfilcon A - (Test Lens) Then Kalifilcon A (Control Lens) | Kalifilcon A - (Control Lens) Then Stenfilcon A - (Test Lens)
Started | 36 | 30
Completed | 36 | 29
Not Completed | 0 | 1
Not completed — Covid-19 related self-isolation | 0 | 1
Period: Second Intervention
Arm/Group | Stenfilcon A - (Test Lens) Then Kalifilcon A (Control Lens) | Kalifilcon A - (Control Lens) Then Stenfilcon A - (Test Lens)
Started | 36 | 29
Completed | 36 | 28
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear test lenses for one week then cross-over to the control lenses for one week.
  stenfilcon A - (Test lens)
  kalifilcon A - (Control Lens)
Arm/Group | Overall Study
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Lens Wettability
Description: Lens wettability on a 0 to 4 descriptive scale, 0.5 steps (0 - Very poor: Immediately displaying non-wetting areas on the lens surface, immediate drying time, 1 - Poor: Irregular surface appearance, drying time << blink time, 2 - Acceptable: Smooth surface appearance immediately after the blink becoming irregular after a while, drying time ≤ blink time, 3 - Good: Typical soft lens appearance with long drying time, 4 - Excellent: Appearance similar to a healthy cornea with very long drying time)
Time Frame: Baseline - after 2 hours of lens wear
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stenfilcon A - (Test Lens): Subjects were randomized to wear test lenses for one week then cross-over to the control lenses for one week.
  stenfilcon A - (Test lens)
- Kalifilcon A - (Control Lens): Subjects were randomized to wear control lenses for one week then cross-over to the test lenses for one week.
  kalifilcon A - (Control lens)
Arm/Group | Stenfilcon A - (Test Lens) | Kalifilcon A - (Control Lens)
Number analyzed (Participants) | 64 | 64
units on a scale | 3.7 (0.4) | 3.7 (0.5)

2. Primary Outcome: Lens Wettability
Description: as for outcome 1
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A - (Test Lens) | Kalifilcon A - (Control Lens)
Number analyzed (Participants) | 64 | 64
units on a scale | 3.5 (0.6) | 3.5 (0.6)

ADVERSE EVENTS:
Time Frame: From dispense up to 1 week on each study lens, a total of 2 weeks
Groups:
- Stenfilcon A - (Test Lens): Subjects were randomized to wear test lenses for one week then cross-over to the control lenses for one week.
- Kalifilcon A - (Control Lens): Subjects were randomized to wear control lenses for one week then cross-over to the test lenses for one week.
Arm/Group | Stenfilcon A - (Test Lens) | Kalifilcon A - (Control Lens)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 1/66 | 0/66
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stenfilcon A - (Test Lens) (N=66) | Kalifilcon A - (Control Lens) (N=66)
Corneal Abrasion (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT04668989/Prot_SAP_000.pdf